CLINICAL TRIAL: NCT03278600
Title: The Value of Tissue-of-origin (ORIGIN-PanCA○R) Profiling in Predicting Primary Site and Directing Therapy in Patients With Cancer of Unknown Primary: a Prospective Randomized Controlled Study
Brief Title: Tissue-of-origin Directing Therapy in Patients With Cancer of Unknown Primary
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xichun Hu, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fudan CUP-001
Record Dates: First submitted 2017-09-08; First posted 2017-09-11 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2021-03

CONDITIONS: Cancer of Unknown Primary Site
MeSH Terms: conditions — Neoplasms, Unknown Primary

STUDY DESIGN:
Intervention Model Description: Tissue-of-origin test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- site-specific therapy (Experimental): standard treatments of sites of origin
  Interventions: Genetic: tissue-of-origin (ORIGIN-PanCA○R) profiling
- standard empiric chemotherapy (Active Comparator): standard empiric chemotherapy
  Interventions: Genetic: tissue-of-origin (ORIGIN-PanCA○R) profiling

INTERVENTIONS:
Genetic: tissue-of-origin (ORIGIN-PanCA○R) profiling — 90-gene assay to predict the primary tumor site

SUMMARY:
This study is designed to evaluate the value of tissue-of-origin (ORIGIN-PanCA○R) profiling in predicting primary site and directing therapy in patients with cancer of unknown primary.

ELIGIBILITY:
Inclusion Criteria:

* had a diagnosis of cancer of unknown primary (CUP) after a standard evaluation (medical history, physical examination, blood counts, chemistry profile, chest/abdomen computed tomography scans, positron emission tomography scan, and directed evaluation of all symptomatic areas). Patients were required to have one of the following histologies: adenocarcinoma, poorly differentiated neoplasms, poorly differentiated carcinoma, squamous carcinoma. Sufficient archived biopsy tissue from a surgical or core needle biopsy was required to perform the molecular profiling assay. Eastern Cooperative Oncology Group performance status of 0 to 2; no previous systemic therapy; measurable or evaluable disease (RECIST); and adequate organ function.

Exclusion Criteria:

* carcinoma limited to single site which can be potentially cured by surgery of radiotherapy.patients with symptomatic brain metastases, active clinical severe infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-03-18 (Actual)

PRIMARY OUTCOMES:
progression free survival | 6 months

SECONDARY OUTCOMES:
overall response rate | 2 months
overall survival | 12 months
Adverse Events | 2 months
biomarker analysis | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Cancer Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu X, Zhang X, Jiang S, Mo M, Wang Q, Wang Y, Zhou L, Hu S, Yang H, Hou Y, Chen Y, Lu X, Wang Y, Zhou X, Li W, Chang C, Yang X, Chen K, Cao J, Xu Q, Sun Y, Luo J, Luo Z, Hu X. Site-specific therapy guided by a 90-gene expression assay versus empirical chemotherapy in patients with cancer of unknown primary (Fudan CUP-001): a randomised controlled trial. Lancet Oncol. 2024 Aug;25(8):1092-1102. doi: 10.1016/S1470-2045(24)00313-9. Epub 2024 Jul 25. PMID 39068945